CLINICAL TRIAL: NCT02735031
Title: Effect of the GLP-1 Receptor Agonist Exenatide on Impaired Hypoglycaemic Awareness in Type 1 Diabetes
Brief Title: Exenatide and Impaired Hypoglycaemic Awareness in Type 1 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESR-15-10862
Record Dates: First submitted 2016-02-22; First posted 2016-04-12 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus, Type 1; Hypoglycemia
Keywords: Glucagon-Like Peptide 1; Impaired hypoglycemic awareness
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXENATIDE (Active Comparator): Exenatide
  * week 1-2: 5 µg twice daily
  * week 3-6: 10 µg twice daily (if tolerated)
  Interventions: Drug: Exenatide
- PLACEBO (Placebo Comparator): Placebo matched to exenatide
  * week 1-2: 5 µg twice daily
  * week 3-6: 10 µg twice daily (if tolerated)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide — 6 weeks treatment with exenatide on top of insulin treatment
  Other Names: Byetta
  Arms: EXENATIDE
Drug: Placebo — 6 weeks treatment with placebo on top of insulin treatment
  Arms: PLACEBO

SUMMARY:
Approximately 25% of patients with type 1 diabetes have lost the capacity to timely detect hypoglycaemia, a condition referred to as impaired hypoglycaemic awareness (IHA) that causes a six-fold higher risk of severe, potentially hazardous, hypoglycaemia. IHA is usually the end-result of a process of habituation to recurrent hypoglycemia that is potentially reversible. Treatment with glucagon-like peptide (GLP)-1 Receptor Agonists (1RAs) in addition to insulin therapy may decrease the incidence of hypoglycaemia in patients with type 1 diabetes. This study will test the hypothesis that treatment with the GLP-1RA, exenatide, added to basal-bolus insulin therapy will improve awareness of hypoglycaemia in patients with type 1 diabetes and IHA. In a randomized doubleblind placebo-controlled cross-over trial, patients will be treated for 6 weeks with exenatide (or placebo), after which hypoglycemic symptoms and counterregulatory hormone responses will be examined during a hyperinsulinemic hypoglycemic glucose clamp study.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes, disease duration >1 year
* Age >18 years, <70 years
* Insulin treatment according to basal-bolus insulin regimen (injections or insulin pump)
* Impaired hypoglycaemic awareness as assessed by a score of 3 or more on the modified Dutch translation of the Clarke questionnaire
* Glycated haemoglobin (HbA1c) ≥42 mmol/mol (6%) and ≤75 mmol/mol (9.0%)
* Ability to provide informed consent

Exclusion Criteria:

* Treatment with incretin-based therapy
* Known intolerance to GLP-1RAs (including allergy)
* Treatment with glucose-modifying or immune-modifying agents, e.g. prednisolon
* Recent history of myocardial infarction or stroke (past year) or laser coagulation for proliferative retinopathy (past 6 months)
* Proliferative retinopathy
* Symptomatic diabetic neuropathy
* Diabetic nephropathy as reflected by albumin-creatinin ratio >30 mmol/mg or estimated Glomerular Filtration Rate (eGFR) <60 ml/min/1.73 m2
* Known heart failure
* History of pancreatitis (acute or chronic) or pancreatic cancer
* Body-mass index >40 kg/m2
* Use of premixed insulin or of long-acting insulin alone
* Total daily insulin dose requirements <20 units unless on pump treatment
* Pregnancy or unwillingness to undertake measures for birth control

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Symptom score in response to insulin-induced hypoglycaemia | 30 minutes
  Measured during hyperinsulinemic hypoglycaemic glucose clamps

SECONDARY OUTCOMES:
Adrenaline response to insulin-induced hypoglycaemia | 30 minutes
  Measured in plasma during hyperinsulinemic hypoglycaemic glucose clamps
Glucagon response to insulin-induced hypoglycaemia | 30 minutes
  Measured in plasma during hyperinsulinemic hypoglycaemic glucose clamps
Time until glycaemic recovery from hypoglycaemia | 1 hour
  Measured during hyperinsulinemic hypoglycaemic glucose clamps
Maximal glucose excursion post-hypoglycaemia | 1 hour
  Measured during hyperinsulinemic hypoglycaemic glucose clamps
Time until glucose peak post-hypoglycaemia | 1 hour
  Measured after hyperinsulinemic hypoglycaemic glucose clamps
Area under the glucose concentration curve post-hypoglycaemia | 1 hour
  Measured after hyperinsulinemic hypoglycaemic glucose clamps
Hunger score post-hypoglycaemia | 1 hour
  Measured after hyperinsulinemic hypoglycaemic glucose clamps
Carbohydrate requirement after recovery from hypoglycaemia | 1 hour
  Measured after hyperinsulinemic hypoglycaemic glucose clamps by showing pictures of various carbohydrate-containing snacks and beverages
Number of severe hypoglycaemic events during follow-up | 16 weeks
Number of nocturnal hypoglycaemic events during follow-up | 16 weeks
Number of any hypoglycaemic events during follow-up | 16 weeks
Number of hypoglycaemic events measured by glucose sensor monitoring | 1 week
  optional (in participants agreeing to wear a continuous glucose sensor for 5 days)
Time spent under hypoglycaemic conditions measured by glucose sensor monitoring | 1 week
  optional (in participants agreeing to wear a continuous glucose sensor for 5 days)
Glucose variability as measured by glucose sensor monitoring | 1 week
  optional (in participants agreeing to wear a continuous glucose sensor for 5 days)

OTHER OUTCOMES:
Pulse rate | 6 weeks
  Measured during hyperinsulinemic hypoglycaemic glucose clamps
Gastrointestinal side effects | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical centre, Nijmegen, Netherlands